CLINICAL TRIAL: NCT03257787
Title: A Pilot Evaluation of Newly Developed Adhesives and How They Are Impacted by Output
Brief Title: Evaluation of the Performance of a New Adhesive Strip
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CP265_15
Record Dates: First submitted 2017-08-18; First posted 2017-08-22 (Actual); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Ileostomy - Stoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test of a new adhesive strip (Experimental): A new adhesive strip has been developed and will be tested in this investigation.
  Interventions: Other: new adhesive strip

INTERVENTIONS:
Other: new adhesive strip — This is a strip made of a newly developed adhesive

SUMMARY:
This study investigates the performance of a new adhesive strip when impacted by output.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent
2. Be at least 18 years of age and have full legal capacity
3. Have had a stoma for more than one year
4. Have intact skin on the area used in the evaluation
5. Has a stoma with a diameter up to (≤) 35 mm
6. Have a peristomal area accessible for application of adhesive strips (assessed by investigating scientist)

Exclusion Criteria:

1 Currently receiving or have within the past 2 month received radio- and/or chemotherapy 2. Currently receiving or have within the past month received topical steroid treatment in the peristomal skin area or systemic steroid (tablet/injection) treatment.

3. Are pregnant or breastfeeding 4. Having dermatological problems in the peristomal or abdominal area (assessed by investigating scientist) 5. Actively participating in other interventional clinical investigations or have previously participated in this investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2017-08-23 (Actual); Study Completion 2017-09-23 (Actual)

PRIMARY OUTCOMES:
Trans epidermal water loss | 8 hours
  The trans epidermal water loss is a measure of the skins barrier function. There is always a loss of water from the skin due to evaporation. However, when the barrier is damaged this evaporation increases. Thus, trans epidermal water loss can be used to assess damage to the skin.

CONTACTS AND LOCATIONS:
Overall Officials: Lene F Nielsen, Principal Investigator — Head of preclinical department
Locations (1):
- Coloplast A/S, Humlebæk, Denmark